CLINICAL TRIAL: NCT02369406
Title: BHP Early Infant Treatment Study: a Clinical Treatment Trial of HIV+ Infants in Botswana
Brief Title: Early Infant HIV Treatment in Botswana
Acronym: EIT
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Ragon Institute of MGH, MIT and Harvard (Other); Brigham and Women's Hospital (Other); Botswana Harvard Health Partnership (Unknown); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Roger Shapiro, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01AI114235 (NIH)
Record Dates: First submitted 2015-02-12; First posted 2015-02-24 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: HIV; Pediatric AIDS
Keywords: Botswana; Immunology; Antiretroviral Therapy
MeSH Terms: interventions — Nevirapine; lopinavir-ritonavir drug combination; Lamivudine; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Antepartum Cohort (Experimental): 40 children who test HIV-positive within 96 hours after birth (antepartum HIV infection) and are able to initiate ART < 7 days after birth. This cohort will include at least 15 children who start ART < 3 days after birth.
  All infants in the antepartum cohort will initiate ART with Nevirapine, Zidovudine, Lamivudine, and later switch to Kaletra, Zidovudine, Lamivudine.
  Interventions: Drug: Nevirapine; Drug: Kaletra; Drug: Lamivudine; Drug: Zidovudine
- Peripartum Cohort (Experimental): 10 children who test HIV-negative within 96 hours after birth but test HIV-positive <57 days after birth (peripartum HIV infection) and who are able to initiate ART <57 days after birth. This cohort will include at least 10 children who start ART < 21 days after birth.
  The majority of infants in the peripartum cohort will be able to start Kaletra, Zidovudine, Lamivudine as their first regimen, but a minority may start Nevirapine, Zidovudine, Lamivudine and then switch to Kaletra, Zidovudine, Lamivudine.
  Interventions: Drug: Nevirapine; Drug: Kaletra; Drug: Lamivudine; Drug: Zidovudine
- Control Cohort (No Intervention): 25 HIV-infected children who initiated ART at later age ranges (30-365 days for antepartum infection, 57-365 days for peripartum infection or for those with unknown timing of infection) will be enrolled for a single visit that will occur between 24 and 36 months of age. These children will serve as a control group for virologic and immunologic comparisons with children in the prospective cohorts.

INTERVENTIONS:
Drug: Nevirapine
  Other Names: NVP
  Arms: Antepartum Cohort; Peripartum Cohort
Drug: Kaletra
  Other Names: LPV/r
  Arms: Antepartum Cohort; Peripartum Cohort
Drug: Lamivudine
  Other Names: 3TC
  Arms: Antepartum Cohort; Peripartum Cohort
Drug: Zidovudine
  Other Names: ZDV
  Arms: Antepartum Cohort; Peripartum Cohort

SUMMARY:
The overall objective of this study is to determine whether very early antiretroviral treatment (ART) initiation in HIV-infected infants limits the seeding of viral reservoirs and maintains immune responses, potentially allowing future periods off ART.

DETAILED DESCRIPTION:
HIV-1 infection during adulthood leads to a stable, long-lasting viral reservoir in CD4 T cells that persists despite suppressive antiretroviral therapy (ART), and is responsible for rapid viral rebound once treatment is stopped in most cases. In neonates, HIV-1 infection occurs at a time when the adaptive immune system is still in development, which may alter the establishment of a long-lasting viral reservoir and offer opportunities to reduce viral persistence through early antiretroviral treatment. Recently, scientific understanding of neonatal HIV infection has been challenged by the description of an infant who tested positive for HIV at birth, was treated with potent combination antiretroviral therapy (ART) within the first 30 hours of life, and achieved long-term remission of HIV infection when ART was stopped approximately 18 months later. Unfortunately, after 2 years off ART, rebound viremia occurred in this child, yet this case raises the provocative question of whether ART initiated within the first days of life for an antepartum infection, or in the first days/weeks of life for a peripartum infection, can prevent the seeding of a long-lasting reservoir of HIV infected cells in some infants (and therefore lead to long periods of HIV remission off ART).

ELIGIBILITY:
Inclusion Criteria (antepartum infection cohort):

1. Mother/guardian ≥18 years of age and able to provide informed consent
2. Gestational age at birth ≥35 weeks
3. Birth weight ≥2000 grams
4. Age is less than 7 days*
5. HIV-infection identified by testing conducted within 96 hours after birth NOTE: HIV-infection is defined as DNA PCR positive on at least one specimen, with confirmation specimen either positive or pending**
6. Ability to initiate ART within 7 days after birth
7. Eligible for ART through the Botswana government program
8. Ability to be followed in BHP clinic for up to 240 weeks from enrollment#
9. Blood samples collected and submitted for real-time safety lab evaluations; results may be pending at the time of entry.

   * At least half of infants in the antepartum cohort must be < 3 days at enrollment, including 3 of the first 6 infants enrolled.

     * Participants will be offered extended follow-up for up to 576 weeks. However, willingness to participate in optional extended follow-up is not an inclusion criterion.

Inclusion Criteria (peripartum infection cohort):

1. Mother/guardian ≥18 years of age and able to provide informed consent
2. Age is greater than 4 days and less than 57 days
3. HIV-negative within 96 hours after birth NOTE: HIV-negative is defined as HIV-negative by DNA PCR on a single specimen or HIV-negative on 2 separate confirmatory specimens following a re-test of an HIV-positive sample
4. HIV-positive between 96 hours and 56 days after birth NOTE: DNA PCR positive on at least one specimen with confirmation specimen either positive or pending repeat draw or result**
5. Ability to initiate ART at enrollment
6. Eligible for ART through the Botswana government program
7. Ability to be followed in BHP clinic for ART for up to 240 weeks after enrollment#
8. Blood samples collected and submitted for real-time safety lab evaluations (results may be pending at the time of entry).

   * An enrolled infant later determined to be HIV uninfected by confirmatory testing will end participation in the study and this enrollment will not be counted against the total number of enrollments planned.

     * Participants will be offered extended follow-up for up to 576 weeks. However, willingness to participate in optional extended follow-up is not an inclusion criterion.

Inclusion Criteria (control group):

1. Mother/guardian ≥18 years of age and able to provide informed consent
2. 24-36 months of age
3. HIV-infection documented within 365 days after birth
4. ART initiated within the following timeframe based on timing of HIV-infection diagnosis > 30-365 days after birth if HIV-infection diagnosed within 96 hours after birth OR > 57-365 days after birth if infant was HIV-negative based on testing performed within 96 hours after birth (or if unknown HIV status < 96 hours from birth) and then found to be HIV-positive based on testing performed between 96 hours and 365 days after birth.
5. After 6 months of ART, no more than one HIV RNA measurement > 400 copies/mL

Exclusion Criteria (for antepartum and peripartum infection cohort):

1. Hospitalization for life-threatening medical illness
2. Medical condition making it unlikely that the infant will survive to 96 weeks
3. If lab values are available prior to enrollment, the following Division of AIDS 2014 graded results, from samples collected within 7 days prior to entry without subsequent testing, will exclude an infant:

   * Grade ≥3 ALT
   * Grade ≥3 AST
   * Grade ≥4 hemoglobin

Note: Baseline lab values may not be available at the time of ART start. However, as soon as these values are available (occasionally within <24 hours), they will be used to make rapid treatment decisions. Neonates with baseline Grade 4 hemoglobin will be called immediately to have ZDV discontinued if the value is confirmed. Neonates with baseline Grade 3 or 4 ALT or AST will be called immediately to stop either NVP or LPV/r if the value is confirmed. Neonates who remain on ART may remain on study. Neonates who discontinue all ART for pre-ART laboratory abnormalities will not be counted against total enrollments.

Exclusion Criteria (control group):

1) < 85% reported adherence to prescribed doses or interruption of ART for more than 7 consecutive days since its initiation.

Ages: 0 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of infants who have treatment-limiting adverse events within the first 14 days of treatment | 14 days
To determine the proportion of infants who fail to achieve at least a 1.5 log10 copies/mL reduction in HIV-1 RNA by the 14th day of treatment | 14 days
To determine the proportion of infants in the antepartum cohort with trough drug concentrations below defined therapeutic ranges at 7 and 14 days of treatment (trough concentrations will be evaluated for NVP, ZDV, 3TC) | 14 days
To evaluate virologic and immunologic outcomes of very early ART in infancy | 84-96 weeks
  Virologic outcomes after early ART: We will evaluate how the timing of HIV infection and the timing of ART initiation affect the size and composition of the viral reservoir over time.
  Immunologic outcomes after early ART: We will evaluate how immune activation and immune activity against HIV-1 contribute to the size and composition of the HIV-1 reservoir over time in infants treated early with suppressive ART.
  Control Group Comparisons. We will evaluate virologic and immunologic outcomes at a single time point in children for whom ART initiation was later than in the prospective cohorts, and compared with immunologic testing of stored specimens from HIV exposed uninfected and HIV unexposed children.

SECONDARY OUTCOMES:
Number of participants with HIV-1 RNA levels <40 copies/mL | up to 576 weeks
Number of participants with reservoir HIV-1 DNA (in copies/million peripheral blood mononuclear cells, PBMCs) below the level of detection for total virus | up to 576 weeks
  Threshold of detection is expected to be approximately 5 copies/million PBMCs, but varies by sample volume available.
Median CD4 cell count (cells/mm3) and 95% confidence intervals among participants | up to 576 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roger L Shapiro, MD, MPH, Principal Investigator — Harvard School of Public Health (HSPH); Daniel R. Kuritzkes, MD, Principal Investigator — Brigham and Women's Hospital; Mathias Lichterfeld, MD, PhD, Principal Investigator — Ragon Institute of MGH, MIT and Harvard
Locations (1):
- Botswana Harvard HIV/AIDS Institute Partnership, Gaborone, Botswana

REFERENCES:
- [Background] Hartana CA, Garcia-Broncano P, Rassadkina Y, Lian X, Jiang C, Einkauf KB, Maswabi K, Ajibola G, Moyo S, Mohammed T, Maphorisa C, Makhema J, Yuki Y, Martin M, Bennett K, Jean-Philippe P, Viard M, Hughes MD, Powis KM, Carrington M, Lockman S, Gao C, Yu XG, Kuritzkes DR, Shapiro R, Lichterfeld M. Immune correlates of HIV-1 reservoir cell decline in early-treated infants. Cell Rep. 2022 Jul 19;40(3):111126. doi: 10.1016/j.celrep.2022.111126. PMID 35858580
- [Background] Ibrahim M, Maswabi K, Ajibola G, Moyo S, Hughes MD, Batlang O, Sakoi M, Auletta-Young C, Vaughan L, Lockman S, Jean-Philippe P, Yu X, Lichterfeld M, Kuritzkes DR, Makhema J, Shapiro RL. Targeted HIV testing at birth supported by low and predictable mother-to-child transmission risk in Botswana. J Int AIDS Soc. 2018 May;21(5):e25111. doi: 10.1002/jia2.25111. PMID 29852062
- [Background] Maswabi K, Ajibola G, Bennett K, Capparelli EV, Jean-Philippe P, Moyo S, Mohammed T, Batlang O, Sakoi M, Lockman S, Makhema J, Lichterfeld M, Kuritzkes DR, Hughes MD, Shapiro RL. Safety and Efficacy of Starting Antiretroviral Therapy in the First Week of Life. Clin Infect Dis. 2021 Feb 1;72(3):388-393. doi: 10.1093/cid/ciaa028. PMID 31927562
- [Background] Garcia-Broncano P, Maddali S, Einkauf KB, Jiang C, Gao C, Chevalier J, Chowdhury FZ, Maswabi K, Ajibola G, Moyo S, Mohammed T, Ncube T, Makhema J, Jean-Philippe P, Yu XG, Powis KM, Lockman S, Kuritzkes DR, Shapiro R, Lichterfeld M. Early antiretroviral therapy in neonates with HIV-1 infection restricts viral reservoir size and induces a distinct innate immune profile. Sci Transl Med. 2019 Nov 27;11(520):eaax7350. doi: 10.1126/scitranslmed.aax7350. PMID 31776292
- [Background] Ajibola G, Garcia-Broncano P, Maswabi K, Bennett K, Hughes MD, Moyo S, Mohammed T, Jean-Philippe P, Sakoi M, Batlang O, Lockman S, Makhema J, Kuritzkes DR, Lichterfeld M, Shapiro RL. Viral Reservoir in Early-Treated Human Immunodeficiency Virus-Infected Children and Markers for Sustained Viral Suppression. Clin Infect Dis. 2021 Aug 16;73(4):e997-e1003. doi: 10.1093/cid/ciab143. PMID 33605999
- [Background] Mistry R, Wilke R, Challiss RA. Modulation of NMDA effects on agonist-stimulated phosphoinositide turnover by memantine in neonatal rat cerebral cortex. Br J Pharmacol. 1995 Feb;114(4):797-804. doi: 10.1111/j.1476-5381.1995.tb13275.x. PMID 7773540
- [Background] Gribakin FG. [Peculiarities of transmission of the receptor signal in photoreceptors]. Zh Evol Biokhim Fiziol. 1981 Sep-Oct;17(5):498-502. Russian. PMID 7293566
- [Background] Helbing C, Gallimore C, Atkinson BG. Characterization of a Rana catesbeiana hsp30 gene and its expression in the liver of this amphibian during both spontaneous and thyroid hormone-induced metamorphosis. Dev Genet. 1996;18(3):223-33. doi: 10.1002/(SICI)1520-6408(1996)18:33.0.CO;2-B. PMID 8631156
- [Background] Ibrahim M, Moyo S, Mohammed T, Mupfumi L, Gaseitsiwe S, Maswabi K, Ajibola G, Gelman R, Batlang O, Sakoi M, Auletta-Young C, Makhema J, Lockman S, Shapiro RL. Brief Report: High Sensitivity and Specificity of the Cepheid Xpert HIV-1 Qualitative Point-of-Care Test Among Newborns in Botswana. J Acquir Immune Defic Syndr. 2017 Aug 15;75(5):e128-e131. doi: 10.1097/QAI.0000000000001384. PMID 28350554
- [Background] Hartana CA, Broncano PG, Maswabi K, Ajibola G, Moyo S, Mohammed T, Maphorisa C, Makhema J, Powis KM, Lockman S, Burbelo PD, Gao C, Yu XG, Kuritzkes DR, Shapiro R, Lichterfeld M. Immune Modulation of HIV-1 Reservoir Size in Early-Treated Neonates. J Infect Dis. 2023 Aug 11;228(3):281-286. doi: 10.1093/infdis/jiad173. PMID 37201510
- [Background] Ajibola G, Maswabi K, Hughes MD, Bennett K, Pretorius-Holme M, Capparelli EV, Jean-Philippe P, Moyo S, Mohammed T, Batlang O, Sakoi M, Ricci L, Lockman S, Makhema J, Kuritzkes DR, Lichterfeld M, Shapiro RL. Brief Report: Long-Term Clinical, Immunologic, and Virologic Outcomes Among Early-Treated Children With HIV in Botswana: A Nonrandomized Controlled Clinical Trial. J Acquir Immune Defic Syndr. 2023 Apr 15;92(5):393-398. doi: 10.1097/QAI.0000000000003147. PMID 36729692
- [Derived] Moraka NO, Garcia-Broncano P, Hu Z, Ajibola G, Bareng OT, Pretorius-Holme M, Maswabi K, Maphorisa C, Mohammed T, Gaseitsiwe S, VanZyl GU, Kuritzkes DR, Lichterfeld M, Moyo S, Shapiro RL. Patterns of pretreatment drug resistance mutations of very early diagnosed and treated infants in Botswana. AIDS. 2021 Dec 1;35(15):2413-2421. doi: 10.1097/QAD.0000000000003041. PMID 34324451